CLINICAL TRIAL: NCT01526564
Title: Phase III Study of Acetyl-L-Carnitine (ALC) Hydrochloride Enteric-coated Tablets in Treatment of Peripheral Sensory Neuropathy in Anti-cancer Chemotherapeutics Induce
Brief Title: Clinical Study on Acetyl-L-Carnitine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZHAOKE-2007L03540
Record Dates: First submitted 2010-09-14; First posted 2012-02-06 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2012-02

CONDITIONS: Peripheral Sensory Neuropathy
Keywords: Chemotherapy-induced peripheral neuropathy (CIPN)
MeSH Terms: interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALC (Active Comparator): ALC
  Interventions: Drug: Acetylcarnitine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylcarnitine — Administration of enteric-coated tablets with warm water at half an hour after meals, 1g (2 tablets) each time, 3 times a day, and the interval at or >4 hours for 8 weeks
  Other Names: NICETILE
  Arms: ALC
Drug: Placebo — 3 t.i.d, two plates per time
  Arms: Placebo

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common clinical dose-limiting adverse drug reaction, and the primary manifestations are different degree of neuromotor, sensorineural and autonomic nervous dysfunction.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled and parallel clinical trial is to observe the efficacy and safety of the Acetyl-L-Carnitine Hydrochloride enteric-coated tablets in treatment of peripheral sensory neuropathy that anti-cancer chemotherapeutics induce.

ELIGIBILITY:
Inclusion Criteria:

* Patients had signed the Informed Consent Form
* Male or Female
* Age 18-75 years old
* Patients who have treated with Taxoids, Satraplatin and Vincristine; The peripheral sensory neuropathy grading after chemotherapy was >/=grade 3 or grade 2 lasting for one month
* The course of neuropathy was </=6 months
* No need to continue chemotherapy according to the condition nor refusing chemotherapy
* At least one of the neuroelectrophysiological examine results were abnormal
* Physical Condition Score (KPS) >/=60
* Anticipated lifetime>/=60.

Exclusion Criteria:

* Patients whose peripheral sensory neuropathy was induced by medicines except of the Taxoids, Satraplatin and vincristine anti-cancer chemotherapeutics
* Diabetics
* Peripheral sensory neuropathy was induced by Vitamin deficiency, infections, trauma, toxicosis, compression, and ischemia
* Peripheral sensory neurologic dysfunction that induced by lesions of central nervous system; hereditary neuropathy
* Patients who have treated by other medicines for peripheral sensory neuropathy in 30 days
* Patients had treated by other clinical trial medicines or participated into other trials in 30 days
* Patients had active infections
* Any clinical problems out of control
* Women in pregnancy and lactation, Subjects with no compliance.

Ages: 18 Weeks to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2008-08; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Changes in peripheral sensory neuropathy grades | Base and eighth week
  Changes in peripheral sensory neuropathy grades after eight weeks treatment

SECONDARY OUTCOMES:
Changes in Neuroelectrophysiological test | Base and eighth week
  Changes in Neuroelectrophysiological test after eight weeks ALC or placebo treatment
Changes in Cancer-related fatigue level | Base and eighth week
  Changes in Cancer-related fatigue level after eigth weeks treatment
Changes in Physical Condition Score | Base and eighth week
  Changes in Physical Condition Score after eight weeks treatment